CLINICAL TRIAL: NCT02032134
Title: Experimental Protocol for the Infusion of Platelets,Cryopreserved With Dimethyl Sulphoxide (DMSO) and Obtained From Multiple Donors Buffy Coats, in Patients With Severe Thrombocytopenia
Brief Title: Protocol for the Infusion of Buffy Coat-derived Cryopreserved Platelets in Patients With Severe Thrombocytopenia
Acronym: MICE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment failure within the interval of available CRY BC-PLTs for the study
Sponsor: Napolitano Mariasanta (Other)
Collaborators: Regione Sicilia (Unknown)
Responsible Party: Sponsor-Investigator, Napolitano Mariasanta, Assistant Professor (ricercatore td), University of Palermo
Organization: University of Palermo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUP: G33F1100003000
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Thrombocytopenia; Primary Thrombocytopenia,Unspecified; Thrombocytopenia Chemotherapy Induced
Keywords: Cryopreserved platelets, thrombocytopenia, DMSO
MeSH Terms: conditions — Thrombocytopenia | interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with severe thrombocytopenia (Other): Intervention Patients with severe thrombocytopenia with an active bleeding, in preparation for surgery, or after chemotherapy (prophylaxis of bleeding),will receive transfusion of Pooled Platelets Cryopreserved In DMSO With a New System
  Interventions: Biological: Transfusion of Pooled Platelets Cryopreserved In DMSO

INTERVENTIONS:
Biological: Transfusion of Pooled Platelets Cryopreserved In DMSO — Patients with severe thrombocytopenia will be admitted as in patients at the Hematology Unit of the Policlinic "P. Giaccone"- Palermo, if they require platelet transfusion (for bleeding, in preparation for surgery, after chemotherapy); they will receive buffy coat derived cryopreserved platelets,after thawing
  Other Names: New Cryopreservation kit (Promedical ®); Buffy Coat Pooled Platelets Cryopreserved In DMSO

SUMMARY:
The increasing need for blood components and the increasingly careful donor selection procedures, make the availability of blood components very reduced, in particular for platelets that are currently administered preferably "fresh" or cryopreserved, only in emergency conditions.

Exceeding this limit through the spread of use of cryopreserved platelets in the common clinical practice, might help clinicians to avoid wasting valuable products and face periods of particular shortage of donors Some studies already published in the literature over the last decade (1,2) have demonstrated the safety and efficacy of autologous cryopreserved platelets .

The main objective of the proposed study is to evaluate the efficacy and safety of platelets, cryopreserved with DMSO using a a new method, in patients with severe thrombocytopenia.

This is the in vivo phase of a study where availability and efficacy of cryopreserved platelets has been assessed in vitro.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the hemostatic efficacy and safety in the recipients of platelets obtained from buffy coat of multiple donors (five), cryopreserved with DMSO using a new patented method, up to 9 months from the collection.

Further goals are the registration of any related- adverse event (idiosyncrasy, allergy, toxicity)

ELIGIBILITY:
Inclusion Criteria:

Cryopreserved buffy coat pooled platelets will be infused, after being thawed, in inpatients at U.O. of Hematology -Policlinic "P. Giaccone"-Palermo, falling into one of the following categories:

* Stable clinical conditions and no complications with platelets ≤ 10,000/microliter;
* With active bleeding and ≤ 20,000 platelets/microliter;
* In the presence of: high blood pressure, high fever, rapid drop in platelets, infection, chemotherapy, coagulation abnormalities with ≤ 20,000 platelets/microliter.

Exclusion Criteria:

Patients

* Suffering from congenital immunodeficiency
* Allogeneic bone marrow transplant candidates
* Bone Marrow Donors for transplantation
* Undergoing bone marrow transplant or
* Suffering from Hodgkin's disease and treated with purine analogues (Fludarabine, cladribine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of infused cryopreserved platelets (changes in platelets count will be determined at 1 hour and 24 hours post-transfusion) | 1 Hour and 24 hours post-transfusion
  To evaluate the availability of cryopreserved platelets after transfusion, the correct count (the number of platelets poured and the body surface, BMI, recipient) of platelets will be determined at 1 hour and 24 hours post transfusion, respectively

SECONDARY OUTCOMES:
Safety of cryopreserved platelets | During transfusion and within 48 hours after transfusion
  Any transfusion-related side effect (i.e. idiosyncrasy, allergy, toxicity) will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Siragusa, MD, Study Director — Hematology Unit- University of Palermo; Mariasanta Napolitano, MD, Principal Investigator — Hematology Unit- University of Palermo
Locations (1):
- AOUP "P.Giaccone"-Hematology Unit, Palermo, Regione Sicilia, Italy

REFERENCES:
- [Background] Wautier JL. Safety and usefulness of autologous cryopreserved platelets. Lancet. 2002 Dec 14;360(9349):1985. doi: 10.1016/S0140-6736(02)11893-9. No abstract available. PMID 12493312
- [Background] Liu GQ, Ding HF, Lu XJ, Xu M, Xing J, Zhao X, Han F, Shang YH. [The efficacy and safety of autologous cryopreserved platelet transfusion in management of thrombocytopenia after chemotherapy in hematological malignancy]. Zhonghua Nei Ke Za Zhi. 2012 Mar;51(3):188-91. Chinese. PMID 22781890
- [Background] Heal JM, Blumberg N. Optimizing platelet transfusion therapy. Blood Rev. 2004 Sep;18(3):149-65. doi: 10.1016/S0268-960X(03)00057-2. PMID 15183900
- [Background] Murphy MF, Brozovic B, Murphy W, Ouwehand W, Waters AH. Guidelines for platelet transfusions. British Committee for Standards in Haematology, Working Party of the Blood Transfusion Task Force. Transfus Med. 1992 Dec;2(4):311-8. doi: 10.1111/j.1365-3148.1992.tb00175.x. PMID 1339584
- [Background] Dumont LJ, Cancelas JA, Dumont DF, Siegel AH, Szczepiorkowski ZM, Rugg N, Pratt PG, Worsham DN, Hartman EL, Dunn SK, O'Leary M, Ransom JH, Michael RA, Macdonald VW. A randomized controlled trial evaluating recovery and survival of 6% dimethyl sulfoxide-frozen autologous platelets in healthy volunteers. Transfusion. 2013 Jan;53(1):128-37. doi: 10.1111/j.1537-2995.2012.03735.x. Epub 2012 Jun 7. PMID 22671278
- [Background] Meyer E, Delaney M, Lin Y, Morris A, Pavenski K, Tinmouth A, Murphy M, Slichter SJ, Heddle N, Dumont LJ. A reporting guideline for clinical platelet transfusion studies from the BEST Collaborative. Transfusion. 2013 Jun;53(6):1328-34. doi: 10.1111/j.1537-2995.2012.03906.x. Epub 2012 Sep 25. PMID 23003345
- [Background] Dumont LJ, Dumont DF, Unger ZM, Siegel A, Szczepiorkowski ZM, Corson JS, Jones MK, Christoffel T, Pellham E, Bailey SL, Slichter SJ; BEST Collaborative. A randomized controlled trial comparing autologous radiolabeled in vivo platelet (PLT) recoveries and survivals of 7-day-stored PLT-rich plasma and buffy coat PLTs from the same subjects. Transfusion. 2011 Jun;51(6):1241-8. doi: 10.1111/j.1537-2995.2010.03007.x. Epub 2011 Jan 7. PMID 21214584
- [Derived] Napolitano M, Mancuso S, Raso S, LoCoco L, Arfo PS, De Francisci G, Dieli F, Caccamo N, Reina A, Dolce A, Agliastro R, Siragusa S. Buffy coat-derived platelets cryopreserved using a new method: Results from a pivotal clinical trial on thrombocytopenic patients with acute leukaemia. Transfus Apher Sci. 2019 Dec;58(6):102666. doi: 10.1016/j.transci.2019.10.008. Epub 2019 Nov 5. PMID 31753773